CLINICAL TRIAL: NCT04078789
Title: Evaluation of the Care Path of Patients Who Have Been Sexually Assaulted, at Raymond Poincaré Hospital (France)
Brief Title: Evaluation of the Care Path of Patients Who Have Been Sexually Assaulted
Acronym: AS UMJ/SMI RPC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190619
Record Dates: First submitted 2019-09-02; First posted 2019-09-06 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Sexually Transmitted Diseases
Keywords: sex offenses; sexually transmitted diseases; traumatic injury
MeSH Terms: conditions — Sexually Transmitted Diseases; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this study is to describe the care pathway of patients presenting in the medico-judicial unit of the Raymond Poincaré Hospital in Garches, France, following a complaint for sexual assault and suggest ways to improvement of the care adapted to the characteristics of the participants.

DETAILED DESCRIPTION:
AS secondary objectives, the study aims to:

* Analyze the population of victims of sexual assault seen in consultation at the medico-judicial unit of Raymond Poincaré Hospital.
* Analyze the decision elements of the initiation of the post-exposure treatment and evaluate them against the recommendations.
* Analyze the data collected on the patients and their follow-up in consultation of infectious disease of the hospital of Garches following a sexual assault.
* Identify obstacles encountered by participants to follow the complete follow-up path.

For this purpose the data collection will be done initially within the forensic unit of Raymond Poincaré Hospital. Then, in a second step, the patients requiring the setting up of a post-exposure treatment, are addressed in the service of infectious diseases. The compilations of the data necessary for the study will then be continued until 3 months after the sexual assault.

For the collection of data, they will be based on the medical records of the victims.

ELIGIBILITY:
Inclusion Criteria:

* People declared being victim of sexual assault;
* Consult at medical-legal unit;
* Judicial requirement.

Exclusion Criteria:

- Absence of judicial requirement.

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Anyone declaring to be a victim of sexual assault and consulting in the medico-legal unit on judicial requisition (minors and adults).
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
post-exposure prophylaxis requirement and surveillance termination | at 1 year
  Prevalence of a consultant victim at the medico-legal unit, requiring post-exposure prophylaxis and completing their post-sexual assault surveillance.

SECONDARY OUTCOMES:
Consulting at the medico-legal unit | at 1 year
  Description of victims consulting at the medico-legal unit.
Follow-up in medico-legal unit | at 1 year
  Follow-up of the start of the post-exposure prophylaxis: indication, difficulty of the prescription, respect of the recommendations.
Follow-up in the infectious diseases department | at 1 year
  Description of the patients followed in the department of acute medicine specializing in infectious diseases sent by the medico-legal unit following sexual assault: monitoring of sexually transmitted infections, aspects of psychological care, state of coverage vaccine, rate of completion, causes of cessation of the treatment, reasons for the failure of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Céline Dufort, MD, Principal Investigator — Unité médico-judiciaire (UMJ), Hôpital Raymond Poincaré, Garches, France; Dhiba Marigot-Outtandy, MD, Study Director — Médecine aiguë spécialisée, Hôpital Raymond Poincaré, Garches, France

IPD SHARING:
Plan to Share IPD: No